CLINICAL TRIAL: NCT00272038
Title: Phase II Study Investigating the Efficacy and Activity of Single Agent Erlotinib in Chemotherapy-Naive Androgen Independent Prostate Cancer
Brief Title: Single Agent Erlotinib in Chemotherapy-naive Androgen Independent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oncology Specialists, S.C. (Other)
Responsible Party: Principal Investigator, Dr. Sigrun Hallmeyer, Sigrun Hallmeyer, MD Director of Research; Chadi Nabhan, MD Principal Investigator, Oncology Specialists, S.C.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSI3652S (0513); NCT00321841 (obsolete NCT alias)
Record Dates: First submitted 2006-01-03; First posted 2006-01-04 (Estimated); Results first posted 2013-10-17 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tarceva (Experimental): Tarceva 150 mg QD
  Interventions: Drug: Tarceva

INTERVENTIONS:
Drug: Tarceva — 150mg QD
  Other Names: erlotinib

SUMMARY:
Objectives to evaluate the activity of Erlotinib in prostate cancer patients who are hormone refractory and androgen independent and have not been exposed to chemotherapy.

DETAILED DESCRIPTION:
This is a phase II open label single center study that evaluates the activity, efficacy, and toxicity of single agent Tarceva in chemotherapy-naive AIPC patients. Patients will receive single agent Tarceva at 150 mg daily without interruption until disease progression, unacceptable toxicity, or investigator's discretion. Eligible patients are those with documented prostate cancer (regardless of Gleason Score) who are considered hormone refractory as defined below. All patients must fail an anti-androgen withdrawal trial if they were already on such therapy. If patients were on LHRH analogues alone, they must fail the addition of an anti-androgen before being classified as hormone refractory. All patients must have adequate organ functions as specified below and have an ECOG performance status of 2 or less. It is hypothesized that 25 patients will be needed to adequately assess the activity of Tarceva in AIPC.

The activity of Tarceva in other malignancies has been demonstrated with dosed ranging from 100 to 150 mg daily. It is acceptable not to interrupt therapy unless toxicity occurs of disease progression is documented. Starting patients at 150 mg daily seems to be the most logical step, but dose reductions will be implemented based on side effects and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Documented prostate cancer regardless of Gleason score
* Patients should be considered hormone refractory and androgen independent. They must fail LHRH analogues, and anti-androgen withdrawal trial.
* Failure is confirmed by an increase in PSA value of 10% or more than the value immediately before, and confirmed by another assessment 2 weeks later.
* Patients have to have measurable disease either biochemically using rising PSA or/and with metastatic disease to the bone or visceral organs.
* Performance status of 2 or less using ECOG scale.· Adequate liver function tests with ALT/AST being < 3x normal, total bilirubin of 1.5 or less, and adequate renal function measured by a creatinine of 2.0 mg/dl or less. Alkaline phosphatase values are never exclusion criteria if it is deemed related to bone metastases.
* Patients need to have adequate bone marrow function. ANC of 1000 or above, Hgb of 9.0 g/dl or above, and platelets of 100,000 or above. If other causes are affecting plts counts such as autoimmune disorders, patients are allowed on study.
* Patients with inadequate bone marrow function that is deemed related to bone marrow involvement with prostate cancer are allowed at the investigator's discretion.
* Patients with other malignancies are allowed as long as there is no evidence of the other malignancy present at entry time, and it has been 3 years or more since the treatment for the other disorder was completed.
* Patients with prior exposure to investigational therapies including vaccines are allowed on this study as long as their last exposure was 4 weeks prior to study entry.Patients with known bone metastases are allowed to receive intravenous bisphosphonates such as aredia or zometa.
* Patients on oral bisphosphonates are also allowed.
* Chemo Naive

Exclusion Criteria:

* Patients with prior exposure to Tarceva
* Patients who have received any prior systemic chemotherapy for prostate cancer. Exposure to chemotherapy for other malignancies is allowed as long as last chemotherapy was completed 3 years prior to study entry.
* Patients with prior malignancies are excluded except for those who have non-melanoma skin cancers or other cancers that are in remission with the last therapy given 3 years prior to enrollment.
* Prior exposure to any form of steroids is allowed and is not considered exclusion criteria.
* Performance status of 3 or above using ECOG scale.
* Known HIV positive status Known CNS involvement with prostate cancer

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2005-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chadi Nabhan, MD, Principal Investigator — Oncology Specialists, SC
Locations (1):
- Oncology Specialists, SC, Park Ridge, Illinois, United States

REFERENCES:
- [Derived] Nabhan C, Lestingi TM, Galvez A, Tolzien K, Kelby SK, Tsarwhas D, Newman S, Bitran JD. Erlotinib has moderate single-agent activity in chemotherapy-naive castration-resistant prostate cancer: final results of a phase II trial. Urology. 2009 Sep;74(3):665-71. doi: 10.1016/j.urology.2009.05.016. Epub 2009 Jul 17. PMID 19616281

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were those who met the criteria of Castration Resistant Prostate Cancer (CRPC)who had not yet received chemotherapy.
Pre-assignment Details: Patients must have had adquate bone marrow function and, Eastern Cooperative Oncology Group (ECOG) <3, and measurable disease.
Groups:
- Tarceva: Tarceva 150 mg orally every day
Period: Overall Study
Arm/Group | Tarceva
Started | 29
Completed | 22
Not Completed | 7
Not completed — withdrew before they received 2 cycles | 7

BASELINE CHARACTERISTICS:
Arm/Group | Tarceva
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 29
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Overall Clinical Benefit of Tarceva in CRPC.
Description: Overall Clinical Benefit = percentage of partial responders (PR)+ the percentage of patients with stable disease (SD). Partial Response (PR) is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum. Stable Disease (SD)is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease, using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0).
Time Frame: 5 years
Measure: Number; unit: percentage of pts w/clinical benefit
Arm/Group | Tarceva
Number analyzed (Participants) | 22
percentage of pts w/clinical benefit | 36

2. Secondary Outcome: Overall Survival
Description: One year survival rate.
Time Frame: during study
Measure: Number; unit: % of partcipants alive at one year
Arm/Group | Tarceva
Number analyzed (Participants) | 22
% of partcipants alive at one year | 58

3. Secondary Outcome: Time to Disease Progression
Description: Patients were evaluated for response biochemically and radiographically at each response assessment. RECIST 1.0 criteria were used for radiographic response. PSA measurement at a central laboratory was used to assess biochemical response. Patients must have had a baseline PSA of 5 ng/ml to be evaluated for PSA response. PSA was measured every 8 weeks.
  For patients with measurable disease radiographically, PSA progression was not considered as having progressive disease. Refer to study publication for details.
Time Frame: 25 months
Population: 29 participants enrolled. only 22 were evaluable, 4 withdrew consent, 2 had rapid PSA increase & 1 had cord compression
Measure: Median (Full Range); unit: months
Arm/Group | Tarceva
Number analyzed (Participants) | 22
months | 2 [1 to NA] — Not all participants experienced progression

ADVERSE EVENTS:
Arm/Group | Tarceva
Serious Adverse Events (participants affected / at risk) | 12/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tarceva (N=29)
Chest Pain (Musculoskeletal and connective tissue disorders) | 1
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Hematuria (Renal and urinary disorders) | 5
Gastro Intestinal Bleed (Gastrointestinal disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Congestive Heart Failure (Cardiac disorders) | 1
Weakness (General disorders) | 2
Involuntary Movement of Hands and Arms (Musculoskeletal and connective tissue disorders) | 1
Dehydration (General disorders) | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Emboli (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Bowel Obstruction (Gastrointestinal disorders) | 1
Decompensation (General disorders) | 1
Spinal Cord Compression (Musculoskeletal and connective tissue disorders) | 1
Cellulitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tarceva (N=29)
Low Creatinine Grade 3 & 4 (Renal and urinary disorders) | 2
Alkaline Phosphatase High Grade 3 & 4 (Blood and lymphatic system disorders) | 2
Fatigue Grade 3 & 4 (General disorders) | 2
Pneumonia Grade 3 & 4 (Infections and infestations) | 2
Rash Grade 3 & 4 (General disorders) | 2
Diarrhea Grade 3 & 4 (Gastrointestinal disorders) | 3
Aspartate Aminotransferase Elevated Grade 1 - 4 (Blood and lymphatic system disorders) | 2
Anemia Grade 1 & 2 (Blood and lymphatic system disorders) | 12
Arthralgia Grade 1 & 2 (Nervous system disorders) | 9
Appetite decreased Grade 1 & 2 (Gastrointestinal disorders) | 15
Anxiety Grade 1 & 2 (Renal and urinary disorders) | 9
Alkaline Phosphatase Increased Grade 1 & 2 (Renal and urinary disorders) | 3
Bruises easily (Vascular disorders) | 5
Calcium Low Grade 1 & 2 (Gastrointestinal disorders) | 6
Constipation Grade 1 & 2 (Gastrointestinal disorders) | 5
Chest Pain Grade 1 & 2 (General disorders) | 4
Chills Grade 1 & 2 (General disorders) | 5
Cough Grade 1 & 2 (Respiratory, thoracic and mediastinal disorders) | 5
Dsynea on Exertion Grade 1 & 2 (Respiratory, thoracic and mediastinal disorders) | 3
Depression Grade 1 & 2 (Psychiatric disorders) | 10
Dehydration Grade 1 - 4 (Gastrointestinal disorders) | 5
Diarrhea Grade 1 & 2 (Gastrointestinal disorders) | 22
Edema Grade 1 & 2 (General disorders) | 4
Fatigue Grade 1 - 4 (General disorders) | 14
Fever Grade 1 & 2 (Infections and infestations) | 4
Fungal Infection Grade 1 & 2 (Infections and infestations) | 3
Gastroesophageal Reflux Disease Grade 1 & 2 (Gastrointestinal disorders) | 4
Hand Foot Syndrome Grade 1 - 4 (Skin and subcutaneous tissue disorders) | 3
Hematuria Grade 1 & 2 (General disorders) | 5
Hemoptesis Grade 1 & 2 (Respiratory, thoracic and mediastinal disorders) | 3
Headache Grade 1 & 2 (Nervous system disorders) | 6
Hot Flashes Grade 1 & 2 (General disorders) | 5
Hives Grade 1 & 2 (Skin and subcutaneous tissue disorders) | 5
Hyperglycemia Grade 1 - 4 (Gastrointestinal disorders) | 6
Infection Grade 1 & 2 (Infections and infestations) | 7
Insomnia Grade 1 & 2 (Psychiatric disorders) | 5
Itching Grade 1 & 2 (Skin and subcutaneous tissue disorders) | 7
Lymphopenia Grade 1 - 4 (Blood and lymphatic system disorders) | 6
Lightheadedness Grade 1 & 2 (Nervous system disorders) | 8
Libido decreased Grade 1 & 2 (General disorders) | 4
Mouth Sores Grade 1 & 2 (Gastrointestinal disorders) | 7
Mouth Dry Grade 1 & 2 (Gastrointestinal disorders) | 11
Nail changes Grade 1 & 2 (Skin and subcutaneous tissue disorders) | 2
Potassium Decreased Grade 1 & 2 (Blood and lymphatic system disorders) | 2
Potassium Increased Grade 1 & 2 (Blood and lymphatic system disorders) | 2
Protein Decreased Grade 1 & 2 (Gastrointestinal disorders) | 2
Renal Insufficiency Grade 1 - 4 (Renal and urinary disorders) | 3
Swallowing Difficulty Grade 1 & 2 (Gastrointestinal disorders) | 2
Sodium Decreased Grade 1 & 2 (Gastrointestinal disorders) | 2
Taste Change Grade 1 & 2 (Gastrointestinal disorders) | 2
Urinary Tract Infection Grade 1 & 2 (Infections and infestations) | 2
Wheezing Grade 1 & 2 (Respiratory, thoracic and mediastinal disorders) | 2
Blood Urea Nitrogen increased Grade 1 & 2 (Renal and urinary disorders) | 2
Creatinine Increased Grade 1 & 2 (Renal and urinary disorders) | 2
Eyes dry Grade 1 & 2 (General disorders) | 2
Eyes Watery Grade 1 & 2 (General disorders) | 2
Memory Loss Grade 1 & 2 (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes